CLINICAL TRIAL: NCT05744050
Title: The Impact of Food Reformulation on Energy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Responsible Party: Principal Investigator, Eric Robinson, Prof., University of Liverpool
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Reformulation study
Record Dates: First submitted 2023-02-10; First posted 2023-02-24 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Diet, Healthy; Eating Behavior; Obesity
MeSH Terms: conditions — Feeding Behavior; Obesity

STUDY DESIGN:
Intervention Model Description: Repeated measures
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low energy density (Experimental): The meal served at lunch time to participants will have a low energy density of ~1.1kcal/g. All other foods are identical across conditions (e.g. snacks, dinner, dessert)
  Interventions: Behavioral: Low energy density lunch
- Medium energy density (Experimental): The meal served at lunch time to participants will have a low energy density of ~1.7kcal/g. All other foods are identical across conditions (e.g. snacks, dinner, dessert)
  Interventions: Behavioral: Medium energy density lunch
- High energy density (Experimental): The meal served at lunch time to participants will have a low energy density of ~3kcal/g. All other foods are identical across conditions (e.g. snacks, dinner, dessert)
  Interventions: Behavioral: High energy density lunch

INTERVENTIONS:
Behavioral: Low energy density lunch — Particpants will be provided with a lunch low in energy density (~1.1kcal/g)
  Arms: Low energy density
Behavioral: Medium energy density lunch — Participants will be provided with a lunch medium in energy density(~1.7kcal/g)
  Arms: Medium energy density
Behavioral: High energy density lunch — Participants will be provided with a lunch high in energy density (~3kcal/g)
  Arms: High energy density

SUMMARY:
Food prepared outside of the home tends to have a high energy content, and high levels of nutrients of concern (sodium, fat, saturated fat and sugar), especially when compared to home-cooked food. A number of studies suggest that when energy density of a food is manipulated it has a linear effect on energy intake, because consumers tend to eat a constant weight of food. However, recent observational research suggested that up to approximately 1.5-2kcal/g, individuals are relatively insensitive to changes in energy density, and there is no indication of compensation through altering meal size. However, upwards of approximately 1.5-2kcal/g, the authors proposed that individuals compensate for increases in energy density by selecting and consuming smaller meal sizes.

The investigators aim to measure participant's consumption (in grams and kilocalories) of three meals at low, medium and high energy densities, and to measure later food intake to observe any evidence of later compensation in response to experimental condition

DETAILED DESCRIPTION:
See attached protocol document.

ELIGIBILITY:
Inclusion Criteria:

* Currently reside in the United Kingdom
* Over the age of 18 years
* Fluent English speaker
* Like the test foods
* Have a BMI between the ranges of 18.5 and 35.

Exclusion Criteria:

* Pregnant/breastfeeding
* Partaking in a fast or other restrictive eating for religious reasons at time of participation
* Currently following a diet
* On medication that affects appetite
* Being a smoker
* Current or historic eating disorder
* Dietary restrictions/intolerances including:

  * Any allergies
  * Vegan/vegetarian
  * Gluten-free
  * Dairy-free
  * Sugar-free

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Acute intake | 30 minutes after intervention administered
  The investigators will observe differences in consumption (g/kcal) when participants are given a meal covertly manipulated to be low, medium or high in energy density.

SECONDARY OUTCOMES:
Later intake | Up to 7 hours after intervention administered
  The investigators will measure later food intake, in order to observe any evidence of later compensation in response to experimental condition.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Robinson, PhD, Principal Investigator — University of Liverpool
Locations (1):
- University of Liverpool, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Study data (anonymised) will be shared on the Open Science Framework (OSF)
Supporting Information: Study Protocol, SAP
Time Frame: On publication, indefinitely
Access Criteria: Open website
URL: https://osf.io/e67xg/

REFERENCES:
- [Derived] Finlay AH, Boyland EJ, Jones A, Langfield T, Bending E, Malhi MS, Robinson E. Passive overconsumption? Limited evidence of compensation in meal size when consuming foods high in energy density: Two randomised crossover experiments. Appetite. 2024 Sep 1;200:107533. doi: 10.1016/j.appet.2024.107533. Epub 2024 Jun 1. PMID 38825014

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT05744050/Prot_SAP_ICF_000.pdf